CLINICAL TRIAL: NCT01057563
Title: IN-PACT CORO INtimal hyPerplasia evAluated by oCT in de Novo COROnary Lesions Treated by Drug-eluting Balloon and Bare-metal Stent
Brief Title: Intimal Hyperplasia Evaluated by Optical Coherence Tomography (OCT) in de Novo Coronary Lesions Treated by Drug-eluting Balloon and Bare-metal Stent
Acronym: IN-PACT CORO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Francesco Burzotta, MD, PhD, Catholic University of Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A/582/CE/2009
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Neointimal hyperplasia; Drug-eluting balloon; Optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMS group (Active Comparator): Patients undergoing PCI with BMS implantation
  Interventions: Device: bare-metal stent (BMS)
- PRE-DEB group (Active Comparator): Patients undergoing PCI with BMS implantation after lesion predilation with DEB
  Interventions: Device: drug (paclitaxel)-eluting balloon (DEB)
- POST-DEB group (Active Comparator): Patients undergoing PCI with BMS implantation followed by postdilation with DEB
  Interventions: Device: Drug (paclitaxel)-eluting balloon (DEB)

INTERVENTIONS:
Device: drug (paclitaxel)-eluting balloon (DEB) — BMS implantation after lesion predilation with DEB
  Arms: PRE-DEB group
Device: bare-metal stent (BMS) — BMS implantation
  Arms: BMS group
Device: Drug (paclitaxel)-eluting balloon (DEB) — BMS implantation followed by post-dilation with DEB
  Arms: POST-DEB group

SUMMARY:
Restenosis due to neointimal hyperplasia causes repeat target vessel revascularization in a relevant number of patients undergoing percutaneous coronary interventions (PCI). Drug-eluting stents (DES) are currently adopted to reduce the rate of restenosis; however, they may increase risk of stent thrombosis.

Experimental data and first clinical experiences showed that inhibition of neointimal hyperplasia may be obtained by local administration of anti-proliferative drugs (like paclitaxel) loaded on the surface of angioplasty balloons. Data on the efficacy of novel coronary drug-eluting balloons (DEBs) are lacking.

Aims of this open label prospective, randomized trial is to evaluate neointimal hyperplasia in patients undergoing bare-metal stent (BMS) implantation alone compared to those receiving additional DEB use and to assess if the technique of DEB use may affect the degree of neointimal hyperplasia.

Neointimal hyperplasia will be assessed by Optical coherence tomography (OCT).

DETAILED DESCRIPTION:
Background. Restenosis due to neointimal hyperplasia causes repeat target vessel revascularization in a relevant number of patients undergoing percutaneous coronary interventions (PCI). Drug-eluting stents (DES) are currently adopted to reduce the rate of restenosis and repeat revascularizations in the majority of cases. However, a known drawback that limits the clinical application of DES technology is the possible increased risk of stent thrombosis, requiring the need of a prolonged dual antiplatelet therapy. Such phenomenon is strongly related to the profound inhibition of stent strut endothelization, that leads to the presence of uncovered stent struts, and to the persistence of polymer molecules which may induce inflammatory reactions in the vessel wall.

Experimental data and first clinical experiences showed that inhibition of neointimal hyperplasia may be obtained by local administration of anti-proliferative drugs (like paclitaxel) loaded on the surface of angioplasty balloons. Accordingly, drug-eluting balloons (DEBs) are a promising tool to prevent restenosis and avoid the undesiderable persistence of polymer molecules of DES in the vessel wall, thus potentially increasing the safety of PCI Data on the efficacy of novel coronary DEBs and on the best technique to use them are lacking.

Optical coherence tomography (OCT), has a resolution of 5-10 μm, 10 times higher than intravascular ultrasound, thus allowing fine characterization of stent strut coverage and apposition and detection of minimal degree of in-stent neointima hyperplasia.

Objective of the study:

* To evaluate the degree of neointimal hyperplasia in patients undergoing bare-metal stent (BMS) implantation alone compared to those receiving additional DEB use.
* To assess if the technique of DEB use (pre-dilation or post-dilation) may affect the degree of neointimal hyperplasia after BMS implantation.

Study Design. Open label prospective randomized trial comparing the degree of neointimal hyperplasia assessed by OCT in patients treated by BMS implantation alone, BMS implantation after DEB predilation or BMS followed by DEB postdilation.

Consecutive patients undergoing BMS implantation and agreeing to enter the study will be randomized 1:1:1 to

1. BMS implantation.
2. BMS implantation after lesion predilation with DEB
3. BMS implantation followed by post-dilation with DEB. Enrolled patients will undergo a 6-month follow up coronary angiography with OCT evaluation of the stented segment. OCT analysis will be performed by an expert OCT analyst (GF) blinded to the treatment assignment.

Study population. 30 subjects.

Procedure Description. In all eligible patients, PCI with BMS implantation will be performed according to the physician standard practice. All patients will be pre-treated with dual antiplatelet therapy.

General considerations on DEB usage. DEB is mainly intended to serve as drug delivery to the vessel wall and should therefore always cover the stenotic area as well as any extended pre-treated (injured) vessel area including the target lesion and any adjacent (prox and distal) portions when these were eventually previously covered by a stent or dilated by a balloon catheter, incidentally or by intention.

DEB length and positioning within the target lesion must be therefore carefully chosen to avoid geographic miss between the DEB and such extended pre-treated vessel area.

1. BMS group procedure:

   * Lesion predilation with an undersized semi-compliant balloon (balloon to artery ratio: 0.5/1).
   * BMS implantation (stent to artery ration: 1.1/1).
   * Post-dilation of the stented segment with a non-compliant balloon at high pressure (16-18 atm)
2. PRE-DEB group procedure:

   1. Pre-dilation

      * Pre-dilatation of the target lesion with an undersized semi-compliant standard PTCA balloon (balloon to artery ratio: 0.5/1)
   2. DEB dilation:

      * DEB diameter and pressure: nominal DEB diameter must be chosen to guarantee full vessel wall contact at a pressure close or slightly higher of the DEB nominal pressure (balloon to artery ratio: 1/1)
      * DEB length: nominal DEB length must exceed 10 mm (5mm per edge) the length of the stent which is planned to be deployed
      * DEB inflation time: 45 seconds
   3. BMS implantation
   4. Post-dilation

      * Post dilatation of the stented segment must be performed with a non-compliant PTCA balloon
      * Balloon diameter: nominal PTCA balloon diameter must be chosen to reach a balloon to stent ratio of 1:1 at high pressure (16-18 atm)
      * Balloon length and positioning: PTCA balloon length should be shorter than the length of the deployed stent . In case of post stent edge residual stenosis post-dilation balloon must fall within are outside the stent (5mm per edge) which was the previously dilated by the DEB
3. POST-DEB group procedure:

   1. Pre-dilation

      * Pre-dilatation of the target lesion must be performed with an undersized semi-compliant standard PTCA balloon (balloon to artery ratio: 0.5/1)
   2. BMS implantation

      * stent to artery ratio: 1.1/1
      * stent length must allow full coverage of the target lesion with a single stent as well as be 10 mm shorter than the DEB which the operator is planning to use next
   3. Post-dilation

      * Post dilatation of the stented segment must be performed with a non-compliant PTCA balloon
      * Balloon diameter: nominal PTCA balloon diameter must be chosen to reach a balloon to stent ratio of 1:1 at high pressure (16-18 atm)
   4. DEB-dilation

      * DEB length and positioning: DEB length must be 10 mm longer than the previously deployed stent (or than the extended pre-treated area in case of former post-dilation outside the stent edges) and centred within such pre-treated length (5mm per edge)
      * DEB inflation time: 45 seconds
      * Balloon to stent ratio: 1.1:1 at a pressure close or slightly higher of the DEB nominal pressure

The result of the procedure will be assessed by 3-dimensional QCA.

Post-procedural management. All patients will undergo cardiac damage markers (Creatin-kinase-MB and Troponin I) assessment before the procedure, 6 hours after PCI and 24 hours after PCI. Thereafter, further blood samples will be performed only if clinically indicated.

After PCI, patients will be given aspirin (75-100 mg/die) life-long and clopidogrel (75 mg/die) for 3 months (according to the on-label prescription for DEB-treated patients).

Follow-up. Clinical follow-up will take place at 1 month (±1 week), 6 months (±2 weeks) and 1 year (±30 days). At 6-month follow-up all patients will undergo a quantitative coronary angiography (3-dimensional QCA) and Optical Coherence Tomography (OCT) study.

OCT analysis. OCT will be performed with the Imaging system M2 (LightLab Imaging Inc., Westford, Massachusetts), capable of a pullback speed of 2 mm/sec and acquisition frame rate of 15.6/sec, using a non-occlusive technique, with continuous intracoronary iso-osmolar contrast injection.

The entire stent length will be assessed and cross sectional images will be analysed every 0.5 mm.

STRUT COVERAGE The struts will be classified as uncovered if a tissue layer on the endoluminal surface is not visible or covered in the presence of visibile tissue between the endoluminal surface and the lumen.

The tissue coverage thickness will be measured in each strut as the distance from the strut endoluminal surface to the lumen. In each cross section analysed, the following parameters will be calculated: the percentage of covered struts (the number of covered struts/ total number of struts), the percentage of uncovered struts (number of uncovered struts/ total number of struts), the tissue coverage thickness (μm), the tissue coverage area (stent area - lumen area) and its percentage (tissue coverage area/stent area X 100); the tissue volume coverage (tissue coverage area x stent length) and its percentage (tissue coverage volume/stent volume X 100). To assess the pattern of coverage, the ratio between the difference of maximum and the minimum tissue thickness/maximum tissue coverage will be calculated in each frame. A ratio close to 1 indicates an asymmetric tissue coverage, on the opposite a ratio close to 0 indicates a symmetric tissue coverage.

INCOMPLETE STENT APPOSITION A single stent strut will be defined with incomplete stent apposition (ISA) when the distance between its endoluminal surface and the vessel wall will be higher than the entire strut thickness. ISA will be considered present if at least one single strut will be incompletely apposed to the vessel wall. In each OCT frame analysed, the number of struts with ISA and the maximum distance from the endoluminal stent strut to the vessel wall will be measured. The percentage of struts with ISA (number of struts with ISA/total number of struts), according to the presence/absence of tissue coverage, will also be reported. A strut will be defined as protruding when the strut will protrude into the lumen relative to the intima between the adjacent strut sections and the distance between its endoluminal surface and the vessel wall will be less than the entire strut thickness and higher than half of strut thickness. The percentage of protruding struts (number of protruding struts/total number of strut X 100) will be reported, according to the presence/absence of tissue coverage.

Sample size calculation and statistical analysis. The primary endpoint is the neointimal area. Secondary endpoints will be the percentage of uncovered struts, the percentage of struts with ISA and the percentage of protruding struts.

This OCT study is a superiority study and it is expected that additional DEB use to BMS implantation will lead to a reduction of the primary endpoint compared to BMS implantation alone.

Few information is available on neointimal proliferation after BMS implantation: two small non randomized studies reported maximal and minimal neointimal thickness (mm) at 7.3 month follow up (first study) and mean neointimal thickness at 8 month follow up (latter study) being > 4 folds higher in the BMS group compared to the rapamycin eluting stent group, although data on neointimal area are not available. A recent randomized study comparing 12 polymer coated rapamycin-eluting stents to 12 non polymer rapamycin eluting stents reported a neointimal area of 0.3 ± 0.2 mm2 in the polymer stent vs 1.2 ± 0.8 mm2in the non polymer stent, thus with a difference of 0.9 (95% CI 0.3-1.4). Based on these findings, we may hypothesize that additional DEB use will yield to a value of neointimal area close to that reported in the non polymer rapamycin eluting stent and that this would correspond to approximately 50% reduction of neointimal area in the BMS group. To detect such difference, 10 patients will be required in each group with a power of 0.9 at a two- sided type I error of 0.05. As we cannot anticipate whether the timing of additional DEB use: pre or post stenting, might have a different effect on the reduction of neointimal hyperplasia, 10 patients will be allocated in a randomized fashion to the predilatation DEB use group, 10 patients to the postdilatation DEB use group and 10 to the BMS group.

ELIGIBILITY:
Ages Eligible for Study: 18 Years and older Genders Eligible for Study: Both (female sex with child-bearing potential excluded) Accepts Healthy Volunteers: No

Inclusion Criteria:

* Non-diabetic patients with a stable coronary artery disease, undergoing elective PCI with BMS
* de novo non-complex lesions (no bifurcation lesions, no chronic total occlusions, no severe calcifications, no moderate-to-severe tortuosities) located in straight coronary segments.
* lesion length ≥10 mm and <25 mm.
* vessel size requiring a single stent with diameter between 3.0 and 3.5mm.

Exclusion Criteria:

Clinical:

* age <18 years or impossibility to give informed consent,
* diabetes mellitus
* female sex with child-bearing potential,
* life expectancy less than 6 months or any condition impeding clinical follow-up (no fixed address, etc),
* significant platelet count alteration (<100,000 cells/mm3 or > 700,000 cells/mm3),
* gastrointestinal bleeding requiring surgery or blood transfusions within 4 previous weeks,
* participation to another study with any investigational device or drug within which is still in the active phase.
* history of clotting pathology, known hypersensitivity to aspirin, heparin, cobalt- chromium, paclitaxel, contrast dye,
* renal failure with creatinine value > 2.5 mg/dl,
* poor cardiac function as defined by left ventricular global ejection fraction ≤ 30%
* acute myocardial infarction within the past 48 hours.
* non ST-elevation acute coronary syndrome

Angiographic:

* left main coronary artery disease,
* lesions in coronary artery bypass grafts,
* no suitable anatomy for OCT scan
* bifurcation lesions, chronic total occlusions, severe calcifications, moderate-to-severe tortuosities
* presence of additional non target lesions requiring treatment, within and outside the target vessel, which are not successfully treated (non target lesions must be treated prior to the target lesion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: Neo-intimal area (mm²). | 6 months post procedure

SECONDARY OUTCOMES:
Secondary Endpoints: - 6m percentage of uncovered struts. - 6m percentage of struts with ISA. - 6m percentage of protruding struts. | 6 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Burzotta, MD, PhD, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Institute of Cardiology, Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Background] Waugh J, Wagstaff AJ. The paclitaxel (TAXUS)-eluting stent: a review of its use in the management of de novo coronary artery lesions. Am J Cardiovasc Drugs. 2004;4(4):257-68. doi: 10.2165/00129784-200404040-00006. PMID 15285700
- [Background] Unverdorben M, Vallbracht C, Cremers B, Heuer H, Hengstenberg C, Maikowski C, Werner GS, Antoni D, Kleber FX, Bocksch W, Leschke M, Ackermann H, Boxberger M, Speck U, Degenhardt R, Scheller B. Paclitaxel-coated balloon catheter versus paclitaxel-coated stent for the treatment of coronary in-stent restenosis. Circulation. 2009 Jun 16;119(23):2986-94. doi: 10.1161/CIRCULATIONAHA.108.839282. Epub 2009 Jun 1. PMID 19487593
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Two year follow-up after treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. Clin Res Cardiol. 2008 Oct;97(10):773-81. doi: 10.1007/s00392-008-0682-5. Epub 2008 Jun 5. PMID 18536865
- [Background] Prati F, Cera M, Ramazzotti V, Imola F, Giudice R, Albertucci M. Safety and feasibility of a new non-occlusive technique for facilitated intracoronary optical coherence tomography (OCT) acquisition in various clinical and anatomical scenarios. EuroIntervention. 2007 Nov;3(3):365-70. doi: 10.4244/eijv3i3a66. PMID 19737719
- [Background] Chen BX, Ma FY, Luo W, Ruan JH, Xie WL, Zhao XZ, Sun SH, Guo XM, Wang F, Tian T, Chu XW. Neointimal coverage of bare-metal and sirolimus-eluting stents evaluated with optical coherence tomography. Heart. 2008 May;94(5):566-70. doi: 10.1136/hrt.2007.118679. PMID 17923466
- [Background] 7. Tatsuya I, Mitsuyasu T, Yoshihiro T. Optical coherence tomography analysis of neointimal stent coverage in sirolimus eluting stents compared with bare metal stents. American College of Cardiology Scientific Sessions 2006. J Am Coll Cardiol 2006;47 Suppl:A2906-73
- [Background] Moore P, Barlis P, Spiro J, Ghimire G, Roughton M, Di Mario C, Wallis W, Ilsley C, Mitchell A, Mason M, Kharbanda R, Vincent P, Sherwin S, Dalby M. A randomized optical coherence tomography study of coronary stent strut coverage and luminal protrusion with rapamycin-eluting stents. JACC Cardiovasc Interv. 2009 May;2(5):437-44. doi: 10.1016/j.jcin.2009.01.010. PMID 19463468
- [Derived] Burzotta F, Brancati MF, Trani C, Pirozzolo G, De Maria G, Leone AM, Niccoli G, Porto I, Prati F, Crea F. Impact of drug-eluting balloon (pre- or post-) dilation on neointima formation in de novo lesions treated by bare-metal stent: the IN-PACT CORO trial. Heart Vessels. 2016 May;31(5):677-86. doi: 10.1007/s00380-015-0671-3. Epub 2015 Apr 12. PMID 25863804
- [Derived] De Maria GL, Porto I, Burzotta F, Brancati MF, Trani C, Pirozzolo G, Leone AM, Niccoli G, Prati F, Crea F. Dual role of circulating endothelial progenitor cells in stent struts endothelialisation and neointimal regrowth: a substudy of the IN-PACT CORO trial. Cardiovasc Revasc Med. 2015 Jan-Feb;16(1):20-6. doi: 10.1016/j.carrev.2014.10.008. Epub 2014 Oct 31. PMID 25465324
- [Derived] Burzotta F, Brancati MF, Trani C, Porto I, Tommasino A, De Maria G, Niccoli G, Leone AM, Coluccia V, Schiavoni G, Crea F. INtimal hyPerplasia evAluated by oCT in de novo COROnary lesions treated by drug-eluting balloon and bare-metal stent (IN-PACT CORO): study protocol for a randomized controlled trial. Trials. 2012 May 6;13:55. doi: 10.1186/1745-6215-13-55. PMID 22559260